CLINICAL TRIAL: NCT03462420
Title: Physiotherapy Program for Managing Adhesive Capsulitis in Patients With Diabetes: A Pilot Randomized Trial
Brief Title: Physiotherapy Program for Managing Adhesive Capsulitis in Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB#111221
Record Dates: First submitted 2018-02-27; First posted 2018-03-12 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Adhesive Capsulitis; Diabetes Mellitus
Keywords: Adhesive capsulitis; Frozen shoulder; Diabetes; Physiotherapy
MeSH Terms: conditions — Bursitis; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT+ walking (Experimental): Participants in this group will be referred to a physical therapy facility according to their preferences and the intervention will be chosen by the treating physical therapist. In addition, participants will be asked to perform free walking at their own pace for 30-45 min, 5 days per week for 6 consecutive weeks and to record their walking date/time on a diary form provided by the research team before commencing the study. Participants in PT+ group will also be provided with accelerometer to accurately estimate their physical activity level.
  Interventions: Other: Physical Therapy program
- Regular PT (Active Comparator): Participants in this group will be referred to a physical therapy facility according to their preferences and the intervention will be chosen by the treating physical therapist. Participants in this group will not be notified about the walking program.
  Interventions: Other: Physical Therapy program

INTERVENTIONS:
Other: Physical Therapy program — The physical therapy program will be chosen by the treating therapist. However, the most common physiotherapy interventions include therapeutic exercises, joint mobilization techniques and electrotherapy.
  Other Names: Exercises

SUMMARY:
This pilot randomized trial will compare the preliminary effect of a regular physiotherapy (PT) program to a regular PT combined with a progressive walking program (PT+) in patients with and without diabetes who have adhesive capsulitis. After signing the consent form, recruited participants will be randomized into either PT group (control) or PT+ group (experimental). Participants in both groups will be referred to a physical therapy facility. The intervention will be chosen by treating physical therapist. In PT+ group, participants will also be asked to perform free walking at their own pace. Outcomes measures for the primary outcome (shoulder functional performance) will be evaluated at baseline and after 6 weeks. Secondary outcomes (shoulder ROM, pain and function, muscle strength, and physical activity level) will be evaluated at baseline, at 3 and 6 weeks, and again at 12 weeks after enrolment. We expect adding a progressive walking program to regular PT will result in better outcomes.

DETAILED DESCRIPTION:
In this pilot randomized clinical trial, participants will be recruited from an Orthopedic clinic at St. Joseph's Health Care Centre via surgeon referrals and from local primary health care clinics via posters advertising the study. Potential participants will be contacted by the research team at Hand and Upper Limb Centre (HULC) to arrange for their initial evaluation and sign a consent form. Participants who agree to participate in this study will be asked to complete 2 outcomes questionnaires (i.e. SPADI, RAPA) and Katz comorbidity scale.

Next, patients will be randomly assigned to one of the two groups: regular Physical Therapy program (PT) or regular PT which add a progressive walking program (PT+). Stratified randomization by diabetic status and sex will be used. All participants will be referred to a physical therapy facility according to their preferences and the intervention will be chosen by the treating physical therapist. In PT+ group, participants will be asked to perform free walking at their own pace for 30-45 min, 5 days per week for 6 consecutive weeks and to record their walking date/time on a diary form provided by the research team before commencing the study. Participants in PT+ group will also be provided with accelerometer to accurately estimate their physical activity level. Outcomes measures for the shoulder functional performance test (primary outcome) will be evaluated at baseline and after 6 weeks. Secondary outcomes (shoulder ROM, pain and function, muscle strength, and physical activity level) will be evaluated at baseline, at 3 and 6 weeks, and again at 12 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with and without diabetes who have adhesive capsulitis

Exclusion Criteria:

* Previous shoulder surgery or dislocation
* Shoulder severe osteoarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change of shoulder performance from baseline to 6 weeks after physiotherapy | At baseline and again after 6 weeks
  This test is based on repeated shoulder movements at waist and eye level, and over head work. The test will be performed using Functional Impairment Test- Hand and Neck/ Shoulder/Arm (FIT-HaNSA) tests.

SECONDARY OUTCOMES:
Shoulder range of motion | at baseline, at 3 and 6 weeks, and again at 12 weeks after enrollment
  Shoulder range of motion in flexion, abduction, and external rotation
Shoulder pain and function | at baseline, at 3 and 6 weeks, and again at 12 weeks after enrollment
  Shoulder pain and function will be assessed using Shoulder Pain and Disability Index (SPADI) questionnaire
Muscle strength | at baseline, at 3 and 6 weeks, and again at 12 weeks after enrollment
  The muscle power of the shoulder flexors and abductors muscles will be assessed
Physical activity level | at baseline, at 3 and 6 weeks, and again at 12 weeks after enrollment
  The level of activity will be assessed using Rapid Assessment of Physical Activity (RAPA) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — Western University, Canada; Kenneth Faber, MD, Study Chair — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zreik NH, Malik RA, Charalambous CP. Adhesive capsulitis of the shoulder and diabetes: a meta-analysis of prevalence. Muscles Ligaments Tendons J. 2016 May 19;6(1):26-34. doi: 10.11138/mltj/2016.6.1.026. eCollection 2016 Jan-Mar. PMID 27331029
- [Background] Hsu CL, Sheu WH. Diabetes and shoulder disorders. J Diabetes Investig. 2016 Sep;7(5):649-51. doi: 10.1111/jdi.12491. Epub 2016 Mar 16. No abstract available. PMID 27182002
- [Background] Laslett LL, Burnet SP, Jones JA, Redmond CL, McNeil JD. Musculoskeletal morbidity: the growing burden of shoulder pain and disability and poor quality of life in diabetic outpatients. Clin Exp Rheumatol. 2007 May-Jun;25(3):422-9. PMID 17631739
- [Background] Marwick TH, Hordern MD, Miller T, Chyun DA, Bertoni AG, Blumenthal RS, Philippides G, Rocchini A; Council on Clinical Cardiology, American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee; Council on Cardiovascular Disease in the Young; Council on Cardiovascular Nursing; Council on Nutrition, Physical Activity, and Metabolism; Interdisciplinary Council on Quality of Care and Outcomes Research. Exercise training for type 2 diabetes mellitus: impact on cardiovascular risk: a scientific statement from the American Heart Association. Circulation. 2009 Jun 30;119(25):3244-62. doi: 10.1161/CIRCULATIONAHA.109.192521. Epub 2009 Jun 8. No abstract available. PMID 19506108